CLINICAL TRIAL: NCT02434666
Title: Safety and Tolerability of CPC-201 in Patients With Dementia of the Alzheimer's Type Long Term Extension Safety Study in Patients With Dementia of the Alzheimer's Type Who Completed Study CPC-001-07
Brief Title: Long Term Extension Safety Study in Patients With Dementia of the Alzheimer's Type Who Completed Study CPC-001-07
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chase Pharmaceuticals Corporation, an affiliate of Allergan plc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPC-001-10
Record Dates: First submitted 2015-04-28; First posted 2015-05-05 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Dementia of the Alzheimer's Type
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CPC-201 (Experimental)
  Interventions: Drug: CPC-201

INTERVENTIONS:
Drug: CPC-201

SUMMARY:
This is a long-term-safety roll-over extension study for a Phase II Study (Protocol CPC-001-07).

DETAILED DESCRIPTION:
This is a long-term-safety roll-over extension study for a Phase II Study (Protocol CPC-001-07). Patients having safely completed the 12-week maintenance phase of Study CPC-001-07 will be eligible for admission. Subjects will remain on their CPC-201 MTD as determined in Study CPC-001-07. The dose of CPC-201 will be increased from 15 mg/day (administered in Study CPC-001-07) to 20mg/day starting on Day1. For those patients who do not tolerate 20mg/day CPC-201, the dose of CPC-201will be decreased to its previously tolerated level of 15mg/day.

This protocol allows to increase patients' MTD of CPC-201, as previously determined in the Phase II Study (CPC-001-07 protocol) by, 5mg or 10mg increment up to a maximum of 60 mg/day starting on Day7 or Month 3 visits of this extension protocol per Investigator's judgment and patient's tolerability.

This extension study is intended to continue for each enrolled patient for up to 6 months unless medically contraindicated. Patients may withdraw from this study at any time. Upon termination of this study, patients will return to their original daily donepezil dose of 10 mg/day and will continue to receive CPC-201 mg/day for one final week.

ELIGIBILITY:
Inclusion Criteria:

1. Have signed an Institutional Review Board (IRB) approved informed consent document indicating that they understand the purpose of and procedures required by the study and are willing to participate in the study and comply with all study procedures and restrictions. Informed consent must be obtained from the patient and/or a designated representative prior to initiating any procedures of the study.
2. Have safely completed 12 week maintenance phase of CPC-001-07 study.

Exclusion Criteria:

1. Renal and hepatic dysfunction with:

   Total Bilirubin: >1.5 x UNL AST: >2.5 x UNL ALT: >2.5 x UNL Serum Creatinine: >1.5 x UNL Creatinine Clearance: <30 mL/min (calculated by Cockcroft and Gault equation)
2. History or presence of myasthenia.
3. ECG findings of:

   Complete Left Bundle Branch Block; Ventricular pacing; 2nd degree or 3rd degree AV block; Atrial fibrillation or atrial flutter; HR <45 or >100; PR >220 msec; or QTcF >450 msec in male, >470 msec in female
4. Patients considered unlikely to co-operate in the study, and/or poor compliance anticipated by the investigator.
5. Any other clinically relevant acute or chronic diseases which could interfere with patients' safety during the trial, or expose them to undue risk, or which could interfere with study objectives.

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-01-08 (Actual); Primary Completion 2016-10-18 (Actual); Study Completion 2016-11-22 (Actual)

PRIMARY OUTCOMES:
safety and tolerability of the maximum tolerated dose (MTD) of CPC-201 (adverse events) | 6 months
  To evaluate the safety labs and adverse events from baseline, during the study and at the end of the study.

SECONDARY OUTCOMES:
safety and tolerability of CPC-201 20mg/day (adverse events) | 6 months
  To evaluate the safety labs and adverse events from baseline, during the study and at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Minako Koga, Study Director — Chase Pharmaceuticals
Locations (5):
- United States (5):
  - Miami Jewish Health Systems, Miami, Florida
  - Quantum Laboratories, Inc. Memory Disorder Center, Pompano Beach, Florida
  - Premiere Research Institute Neuroscience, West Palm Beach, Florida
  - IU School of Medicine IU Health Neuroscience Center, Indianapolis, Indiana
  - Giles Cromwell, MD, Winston-Salem, North Carolina